CLINICAL TRIAL: NCT00198133
Title: Phase II Study of Alimta (Pemetrexed) Treatment of Advanced Thymoma and Thymic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Joseph Loehrer Sr. (Other)
Responsible Party: Sponsor-Investigator, Patrick Joseph Loehrer Sr., Professor of Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0412-18; IUCRO-0088; IUCRO-0088
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Thymoma; Thymic Carcinoma
Keywords: Thymoma; Thymic Carcinoma
MeSH Terms: conditions — Thymoma | interventions — Pemetrexed

ARMS (1):
- Pemetrexed (Experimental): Pemetrexed infusion once every 21 days (one cycle).
  Interventions: Drug: Premetrexed (Alimta)

INTERVENTIONS:
Drug: Premetrexed (Alimta) — Pemetrexed will be 500 mg/m2 IV every 3 weeks

SUMMARY:
To study the efficacy of Alimta as a single agent in thymic cancers

DETAILED DESCRIPTION:
The broad range of clinical activity of thymic carcinomas makes the likelihood of detecting efficacy of a single agent such as premetrexed a reasonable objective since these malignancies are relatively slow growing and exhibit a broad range of chemosensitivity to antineoplastic agents.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive, recurrent or metastatic thymoma or thymic carcinoma not amenable to potentially curative therapy by surgery. Original biopsy of tumor is sufficient for diagnoses unless otherwise clinically indicated.
* Patients must have measurable disease with at least one bidimensional measurable lesion. Any scans or x-rays used to document measurable disease must be obtained with 6 weeks prior to registration.
* Patients may have had prior chemotherapy for metastatic disease
* Adequate organ function as defined by: bili </=1.5; calc. crt clr of >/=45; hematologic-granulocytes >/=1500 & plt >/=100K.
* Patients who are receiving a stable dose of corticosteroids for myasthenia gravis are eligible.
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Acute intercurrent infection or complications
* pregnancy or lactating patients
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents for a 5-day period (8-day period for long-acting agents.
* Presence of clinically relevant third-space fluid collections that cannot be controlled by a procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Loehrer, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Gbolahan OB, Porter RF, Salter JT, Yiannoutsos C, Burns M, Chiorean EG, Loehrer PJ Sr. A Phase II Study of Pemetrexed in Patients with Recurrent Thymoma and Thymic Carcinoma. J Thorac Oncol. 2018 Dec;13(12):1940-1948. doi: 10.1016/j.jtho.2018.07.094. Epub 2018 Aug 16. PMID 30121390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on getting 27 evaluable patients through a two-stage design
Groups:
- Thymoma: Patients with Thymoma who received Pemetrexed 500 mg/m2 IV every 3 weeks
- Thymic Carcinoma: Patients with Thymic Carcinoma who received Pemetrexed 500 mg/m2 IV every 3 weeks
Period: Overall Study
Arm/Group | Thymoma | Thymic Carcinoma
Started | 16 | 11
Completed | 11 | 3
Not Completed | 5 | 8
Not completed — Disease progression | 2 | 5
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thymoma | Thymic Carcinoma | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (14.2) | 53.3 (14.4) | 53.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 11 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 13 | 10 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete and Partial Response)
Description: The percent of patients having an objective response (complete or partial response) will be estimated with a 95% exact binomial confidence interval for the percent of patients receiving drug. RECIST v1.0 will be used. At least a 30% decrease in the sum of the longest diameter of target lesions in reference to the baseline longest diameter will need to take place to be considered an objective response.
Time Frame: Up to 3 years
Population: All patients with at least one post baseline measurement. (26 evaluable - 15 T and 11 TC patients)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 15 | 11
percentage of participants | 26.7 [7.8 to 55.1] | 9.1 [0.2 to 41.3]

2. Secondary Outcome: Duration of Remission
Description: Will be examined using Kaplan-Meier estimates. Time from earliest confirmed remission criteria until death or progression will be calculated. If a patient continued to be in remission at the end of the study, they will be censored at their last evaluation in the analysis.
Time Frame: Time from the date of remission until progression or death, assessed up to 3 years
Population: All patients with at least one post baseline measurement who had a response of CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 4 | 1
months | 4.0 [3.3 to 6.3] | 3.8 [NA to NA] — Since there was only one patient with an objective response, the confidence interval was not estimable.

3. Secondary Outcome: Grade 3/4 Treatment Related Adverse Events
Description: To determine the toxicity of premetrexed in this patient population, the number of patients who experienced grade 3 or 4 adverse events will be reported that were treatment related (possibly, probably, definitely).
Time Frame: Up to 3 years
Population: All patients enrolled and received treatment
Measure: Number; unit: participants
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 16 | 11
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Beginning of treatment until the end of the study, up to 3 years
Arm/Group | Thymoma | Thymic Carcinoma
Serious Adverse Events (participants affected / at risk) | 2/16 | 3/11
Other Adverse Events (participants affected / at risk) | 16/16 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoma (N=16) | Thymic Carcinoma (N=11)
SUPERIOR VENA CAVA SYNDROME (SVC) (Cardiac disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
DYSPNEA (Gastrointestinal disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
FEVER (General disorders) | 0 | 1
BLOOD INFECTION (STAPHLOCOCCUS HOMINIS) (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
ACHALASIA (Musculoskeletal and connective tissue disorders) | 1 | 0
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoma (N=16) | Thymic Carcinoma (N=11)
ANC (NEUTROPENIA) (Blood and lymphatic system disorders) | 1 | 0
ANEMIA (Blood and lymphatic system disorders) | 0 | 1
ANKLE EDEMA (Blood and lymphatic system disorders) | 0 | 2
BILATERAL ANKLE EDEMA (Blood and lymphatic system disorders) | 1 | 0
EDEMA +1 (Blood and lymphatic system disorders) | 0 | 1
EDEMA - ANKLES (Blood and lymphatic system disorders) | 1 | 0
EDEMA-LEFT ARM (Blood and lymphatic system disorders) | 1 | 0
SWOLLEN FACE/RED (Blood and lymphatic system disorders) | 1 | 0
ARRHYTHIA (TACHYCARDIA) (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
PERICARDIAL TAMPONADE (Cardiac disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 0
DIABETES (Endocrine disorders) | 0 | 1
HYPOTHYROID (Endocrine disorders) | 1 | 0
HYPOTHYROIDISM (Endocrine disorders) | 1 | 1
BLURRY VISION (Eye disorders) | 1 | 0
DRY EYES (Eye disorders) | 0 | 2
EYE DRAINAGE/ REDNESS (Eye disorders) | 1 | 0
EYE SWELLING (Eye disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
ANOREXIA (INTERMITTENT) (Gastrointestinal disorders) | 1 | 0
BLOATING (Gastrointestinal disorders) | 0 | 1
CANDIDA ESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 4 | 6
DIARRHEA (Gastrointestinal disorders) | 5 | 1
DIARRHEA (INTERMITTENT) (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 4 | 2
DYSPEPSIA (HEARTBURN)/REFLUX (Gastrointestinal disorders) | 0 | 1
DYSPEPSIA (INTERMITTENT) (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (STOMACH ACHE) (Gastrointestinal disorders) | 1 | 0
DYSPNEA (Gastrointestinal disorders) | 9 | 8
DYSPNEA (INTERMITTENT) (Gastrointestinal disorders) | 1 | 1
GAS (Gastrointestinal disorders) | 1 | 0
GERD (Gastrointestinal disorders) | 1 | 1
HEARTBURN (Gastrointestinal disorders) | 0 | 1
INCONTINENCE (Gastrointestinal disorders) | 2 | 0
INTEMITTENT DYSPEPSIA (Gastrointestinal disorders) | 0 | 1
INTERMITTENT CONSTIPATION (Gastrointestinal disorders) | 1 | 0
INTERMITTENT DIARRHEA (Gastrointestinal disorders) | 1 | 0
INTERMITTENT DYSPEPSIA (Gastrointestinal disorders) | 2 | 0
INTERMITTENT NAUSEA (Gastrointestinal disorders) | 3 | 2
INTERMITTENT STOMACH PAIN (Gastrointestinal disorders) | 1 | 0
INTERMITTENT VOMITTING (Gastrointestinal disorders) | 1 | 1
MUCOSITIS (Gastrointestinal disorders) | 5 | 0
MUCOSITIS (THRUSH) (Gastrointestinal disorders) | 1 | 0
MUCOSITIS - ORAL CAVITY (MOUTH ULCERS) (Gastrointestinal disorders) | 1 | 0
MUCOSITIS/STOMATITIS (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 6
NAUSEA (INTERMITTENT) (Gastrointestinal disorders) | 2 | 0
NAUSEA INTERMITTENT (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 0
TASTE ALTERATION (Gastrointestinal disorders) | 4 | 2
VOMITING (Gastrointestinal disorders) | 2 | 4
FATIGUE (General disorders) | 12 | 10
FEVER (General disorders) | 3 | 2
INSOMNIA (General disorders) | 8 | 5
INTERMITTENT ARTHRALGIA (General disorders) | 1 | 0
INTERMITTENT CHEST PAIN (General disorders) | 1 | 0
INTERMITTENT INSOMNIA (General disorders) | 1 | 0
INTERMITTENT MIGRAINES (General disorders) | 1 | 0
INTERMITTENT SORE THROAT (General disorders) | 1 | 0
JOINT PAIN (General disorders) | 1 | 0
LEFT SHOULDER PAIN (General disorders) | 0 | 1
LIMBIC ENCEPHALITIS (CHARACTERIZED BY DROWSINESS, HALLUCINATIONS, LOSS OF SHORT TERM MEMORY, CONFUSI (General disorders) | 1 | 0
LT SHOULDER PAIN (General disorders) | 0 | 1
MUSCULOSKELATAL CHEST PAIN (General disorders) | 0 | 1
NIGHT SWEATS (General disorders) | 1 | 1
PAIN (CHEST) (General disorders) | 1 | 0
PAIN - RIGHT CHEST INCISIONAL (General disorders) | 0 | 1
PAIN - RIGHT LUNG (General disorders) | 1 | 0
PAIN - RIGHT SHOULDER (General disorders) | 0 | 1
PAIN - RIGHT UPPER CHEST (General disorders) | 1 | 0
PANIC ATTACK INTERMITENT (General disorders) | 1 | 0
RIGHT HIP PAIN (General disorders) | 0 | 1
RIGHT SHOULDER AND BACK PAIN (General disorders) | 0 | 1
RIGHT-SIDED CHEST PAIN (General disorders) | 0 | 1
RUNNING NOSE (General disorders) | 2 | 0
RUNNY NOSE (General disorders) | 1 | 0
SHOULDER PAIN (General disorders) | 1 | 0
SINUS CONGESTION (General disorders) | 1 | 0
SINUS DRAINAGE (General disorders) | 2 | 1
SORE THROAT (General disorders) | 4 | 0
STOMACH PAIN (General disorders) | 2 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
FLUSHING (INTERMITTENT) (Infections and infestations) | 1 | 0
FUNGAL INFECTION ON ANKLES (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 1 | 0
PHARGNGITIS (Infections and infestations) | 1 | 0
SINUS INFECTIN (Infections and infestations) | 1 | 0
SINUS INFECTION (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 0
SINUSITIS (SINUS INFECTION) (Infections and infestations) | 1 | 0
STAPH INFECTION (Infections and infestations) | 1 | 0
STREP INFLUENZA (Infections and infestations) | 1 | 0
ELEVATED AST (Investigations) | 1 | 0
ELEVATED LFT'S (Investigations) | 1 | 0
ELEVATED LIVER ENZYMES (Investigations) | 0 | 1
ELEVATED LIVER FUNC. TEST (Investigations) | 1 | 0
ELEVATED LIVER FUNCTION TEST (Investigations) | 2 | 0
HYPERBILIRUBINEMIA (Investigations) | 1 | 0
HYPERBILRUBEMIA (Investigations) | 1 | 0
HYPERGLYCEMIA (Investigations) | 0 | 1
HYPERLIPIDEMIA (Investigations) | 0 | 1
ANOREXIA (Metabolism and nutrition disorders) | 7 | 6
ANKLE/KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
ARTHRITIC PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
BACK PAIN (INTERMITTENT FOR YEARS) (Musculoskeletal and connective tissue disorders) | 1 | 0
BONE PAIN (LEGS) (Musculoskeletal and connective tissue disorders) | 0 | 1
CHEST PAIN (MUSCULOSKELATAL) (Musculoskeletal and connective tissue disorders) | 1 | 0
CHEST TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
CYST ON LEFT BUTTOCK (Musculoskeletal and connective tissue disorders) | 1 | 0
GOUT (Musculoskeletal and connective tissue disorders) | 0 | 1
HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN - BACK MIDDLE (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN - HANDS - INTERMITTAT BURNING SENSATION (Musculoskeletal and connective tissue disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 2 | 0
HEADACHES (Nervous system disorders) | 1 | 1
HEADACHES - INTERMITTENT (Nervous system disorders) | 1 | 0
INTERMITTENT TINGLING IN FINGERS AND TOES (Nervous system disorders) | 1 | 0
LEG WEAKNESS (Nervous system disorders) | 0 | 1
NEUROPATHY (Nervous system disorders) | 1 | 0
NEUROPATHY (FEET, TOES, & ELBOW NUMB) (Nervous system disorders) | 0 | 1
NEUROPATHY (FINGERTIPS) (Nervous system disorders) | 1 | 0
NEUROPATHY - FINGERS (Nervous system disorders) | 2 | 1
NEUROPATHY - FINGERS AND TOES (Nervous system disorders) | 1 | 0
NEUROPATHY - HANDS (Nervous system disorders) | 1 | 0
NEUROPATHY - TOES (Nervous system disorders) | 0 | 1
NEUROPATHY, SENSORY: TOES (Nervous system disorders) | 1 | 0
NEUROPATHY-SENSORY- BALL OF FEET (Nervous system disorders) | 0 | 1
NUMBNESS - FEET (Nervous system disorders) | 1 | 0
NUMBNESS - LEFT CHEST INCISIONAL (Nervous system disorders) | 0 | 1
NUMBNESS OF BOTH LEGS (Nervous system disorders) | 1 | 0
RIGHT FOOT TREMOR (Nervous system disorders) | 1 | 0
RIGHT HAND TREMOR (Nervous system disorders) | 1 | 0
SENSORY NEUROPATHY - BOTTOM OF FEET NUMB (Nervous system disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 5 | 2
ANXIETY (INTERMITTENT) (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
IRRITIABLE (Psychiatric disorders) | 1 | 0
MOOD - DEPRESSION (Psychiatric disorders) | 1 | 0
NOCTURIA (Renal and urinary disorders) | 2 | 1
PAIN - KIDNEY AREA LEFT AND RIGHT (Renal and urinary disorders) | 1 | 0
POLYURIA (Renal and urinary disorders) | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0
ASTHMA (BRONCHIOSPASM) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATCLECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 | 6
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
INTERMITTENT HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 2
ALOPECIA - THINNING (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS BILATERALLY (Skin and subcutaneous tissue disorders) | 0 | 1
HIVES (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERPIGMENTATION OF PALMS OF HANDS (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITIUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 1
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 3 | 2
PRURITUS/ITCHING (INTERMITTENT) (Skin and subcutaneous tissue disorders) | 2 | 0
RASH (Skin and subcutaneous tissue disorders) | 6 | 1
RASH (INFUSION SITE) (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (INTERMITTENT) (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (LEFT CHEST) (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (NECK) INTERMITTENT (Skin and subcutaneous tissue disorders) | 1 | 0
RASH - NECK AND ABDOMEN AREA (Skin and subcutaneous tissue disorders) | 0 | 1
RASH - RED FACE AND ARMS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN - RED, RAISED RASH ON NECK AND UPPER CHEST (Skin and subcutaneous tissue disorders) | 0 | 1
SURGERY (REMOVAL SKIN CANCER) FACE & RIGHT ARM (Skin and subcutaneous tissue disorders) | 0 | 1
UPPER CHEST ITCHING (Skin and subcutaneous tissue disorders) | 0 | 1
BLOOD CLOT-LEFT ARM (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1
INTERMITTENT BLOODY NOSE (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes